CLINICAL TRIAL: NCT02377466
Title: Randomized, Double-blind, Multicenter, Phase III Study Comparing the Efficacy and Safety of Retosiban Versus Placebo for Women in Spontaneous Preterm Labor
Brief Title: A Phase III Efficacy and Safety Study of Intravenous Retosiban Versus Placebo for Women in Spontaneous Preterm Labor
Acronym: NEWBORN-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Asset terminated by PIB
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200719; 2014-003326-41 (EudraCT Number)
Record Dates: First submitted 2015-02-26; First posted 2015-03-03 (Estimated); Results first posted 2018-07-19 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Obstetric Labour, Premature
Keywords: Spontaneous Preterm Labor; GSK221149; Retosiban
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Retosiban (Experimental): Retosiban treatment will be administered as a 6 mg IV loading dose over 5 minutes followed by a 6 milligram per hour (mg/hour) continuous infusion over 48 hours. For subjects with an inadequate response after the first hour of treatment, another 6 mg loading dose will be administered and infusion rate will be increased to 12 mg/hour for the remainder of the 48 hour treatment period. The retosiban dosing regimen will require adjustment in subjects treated concomitantly with drugs that are strong Cytochrome 3A4 inhibitors or inducers.
  Interventions: Drug: Retosiban IV infusion
- Placebo (Placebo Comparator): The placebo control will be a normal saline (0.9% sodium chloride [NaCl]) infusion matched for the loading dose and continuous infusion rates, including a dose increase in subjects with an inadequate response after the first hour of treatment.
  Interventions: Drug: Placebo IV infusion

INTERVENTIONS:
Drug: Retosiban IV infusion — Retosiban for IV administration will be supplied as solution for infusion, consisting of a clear colorless solution of retosiban at a concentration of 15 milligram per milliliter (mg/mL).
  Arms: Retosiban
Drug: Placebo IV infusion — 0.9% NaCl matched for the retosiban loading dose and continuous infusion rates
  Arms: Placebo

SUMMARY:
The study's primary objective is to demonstrate the superiority of retosiban to prolong pregnancy and improve neonatal outcomes compared with placebo. It is a Phase III, randomized, double-blind, parallel-group, multicenter study and will be conducted in approximately 900 females, aged 12 to 45 years, with an uncomplicated, singleton pregnancy and intact membranes in preterm labor between 24^0/7 and 33^6/7 weeks of gestation. Eligible maternal subjects will be randomly assigned in a 1:1 ratio to receive either retosiban IV infusion or placebo IV infusion over 48 hours. If not previously administered, antenatal corticosteroid treatment should be administered as either (1) two 12-mg doses of betamethasone given intramuscularly 24 hours apart or (2) four 6-mg doses of betamethasone administered intramuscularly every 12 hours. A single rescue course of antenatal corticosteroids is permitted if the antecedent treatment was at least 7 days prior to study enrolment. Investigators have discretion to use a standardized regimen of magnesium sulphate, as well as intrapartum antibiotic prophylaxis for perinatal group B streptococcal infection. Prior to randomization, each subject will be stratified by progesterone treatment and gestational age. The progesterone strata will consist of subjects on established progesterone therapy or subjects not on established progesterone therapy at Screening. The study will comprise 6 phases: Screening, Inpatient Randomized Treatment, Post Infusion Assessment, Delivery, Maternal Post-Delivery Assessment, and Neonatal Medical Review. The duration of any subject's (maternal or neonatal) participation in the study will be variable and dependent on gestational ages (GA) at study entry and the date of delivery.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent is required prior to a subject's participation in the study and the performance of any protocol specific procedures. Adolescents aged 12 to 17 years must provide written agreement to participate in the study in accordance with applicable regulatory and country or state requirements. Subjects will also be asked to sign a release for medical records at the time of consenting to allow access to both the maternal and neonatal records including information about delivery and infant care as well as information collected prior to the consent having been signed.
* Females aged 12 to 45 years, with an uncomplicated, singleton pregnancy and intact membranes in preterm.
* Gestational age between 24 and 33 weeks as determined by (1) known fertilization date, either in vitro fertilization or intrauterine insemination, (2) last menstrual period confirmed by the earliest ultrasound prior to 24 weeks gestation, or (3) the earliest ultrasound alone prior to 24 weeks gestation, whichever is the most accurate method available for each subject. In situations where prenatal ultrasound records are not available at the time the subject presents, the investigator will make every effort to obtain these records (either via computer records, directly from the subject's primary care obstetrician, or via telephone). However, in cases in which these records are not readily available (e.g., off hours, holiday), it is within the investigator's discretion to use GA based on a verbal history from the subject with the intent of getting confirmation from the medical records as soon as possible.
* Females must be diagnosed with preterm labor according to both of the following criteria: a) Regular uterine contractions at a rate of >=4 contractions of at least 30 seconds' duration during a 30-minute interval confirmed by tocodynamometry and at least 1 of the following, b) Cervical dilation >=2 centimeter (cm) and <=4 cm by digital cervical examination or c) If <2 cm dilation by digital cervical examination, a cervical change consisting of an increase of at least 25% effacement or 1-cm dilation.
* Current or past tocolytic treatment as follows: a) Subjects in whom tocolytic treatment has not been initiated prior to consent are eligible for the study, b) Transferred or referred subjects for whom parenteral magnesium sulfate treatment has been started before Screening are eligible provided they meet all eligibility criteria, c) Subjects receiving a prohibited tocolytic in this study are eligible only if the treatment is stopped before randomization and provided they meet all eligibility criteria, d) Subjects with a historical failure of a tocolytic treatment in a previous episode of preterm labor during the current pregnancy are eligible provided they meet all eligibility criteria.

Exclusion Criteria:

* Fever with a temperature >100.4 degree Fahrenheit (38 degree centigrade) for more than 1 hour or >=101 degree Fahrenheit (38.3 degree centigrade) in the 24 hours prior to the start of study treatment.
* Women with maternal-fetal conditions that potentially necessitate the need for delivery, such as pre-eclampsia or fetal compromise.
* A fetus with any diagnosis, condition, treatment, or other factor that in the opinion of the investigator has the potential to affect or confound assessments of efficacy or safety (for example: nonreassuring fetal status, intrauterine growth restriction, major congenital anomaly).
* Preterm premature rupture of membranes.
* Women with any confirmed or suspected contraindication to prolongation of pregnancy, such as placental abruption, chorioamnionitis, or placenta previa.
* Evidence of polyhydramnios (AFI >25 cm) or oligohydramnios (AFI <5 cm).
* Women with co-morbid medical or obstetric conditions that in the opinion of the investigator have the potential to complicate the pregnancy course and outcomes, such as uncontrolled hypertension or uncontrolled diabetes (if known, history of glycosylated hemoglobin >8% at any time during pregnancy), or compromise the safety of the subject, such as underlying cardiovascular disorder (specifically ischemic cardiac disease, congenital heart disease, pulmonary hypertension, valvular heart disease, arrhythmias, and cardiomyopathy).
* Women with a history of substance abuse during the pregnancy or urine drug screen positive for cocaine, phencyclidine (PCP), methamphetamine, or amphetamine.
* Women in whom the combination of history and screening test results is suggestive of abuse or dependency that may have the potential to complicate the pregnancy outcome.
* Women with any diagnosis, condition, treatment, or other factor that, in the opinion of the investigator, has the potential to affect or confound assessments of efficacy or safety.
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
* History of sensitivity to any of the investigational products (IPs) or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline/ Pharmaceutical Product Development (GSK/PPD) medical monitor, contraindicates the subject's participation.

Ages: 12 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2017-07-24 (Actual); Study Completion 2017-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (46):
- United States (32):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Colton, California
  - GSK Investigational Site, Orange, California
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Columbus, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Maywood, Illinois
  - GSK Investigational Site, Park Ridge, Illinois
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Louisville, Kentucky
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Jackson, Mississippi
  - GSK Investigational Site, Richmond Heights, Missouri
  - GSK Investigational Site, Neptune City, New Jersey
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, The Bronx, New York
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Lancaster, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Tacoma, Washington
- GSK Investigational Site, London, Ontario, Canada
- Italy (2):
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Milan, Lombardy
- Japan (10):
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Miyazaki
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Okinawa
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tochigi
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20387

RESULTS

PARTICIPANT FLOW:
Recruitment Details: NEWBORN-1 was a randomized, double-blind, placebo-controlled, parallel-group, multicenter study to investigate efficacy and safety of retosiban in female participants aged 12 to 45 years with an uncomplicated singleton pregnancy in preterm labor with intact membranes between 24 0/7 and 33 6/7 weeks gestation. The study was conducted in 3 countries.
Pre-assignment Details: Twenty-five participants were randomly assigned to study treatments: 12 participants to retosiban intravenous (IV) infusion and 13 participants to matched placebo IV infusion. Two participants randomized to retosiban arm did not receive study treatment. The study was terminated early due to feasibility of recruiting the study in a timely manner.
Groups:
- Placebo: Placebo was 0.9 percent sodium chloride infusion matched for retosiban volume, IV loading dose over 5 minutes and continuous infusion rate including dose increase in participants with an inadequate response any time after first hour of treatment.
- Retosiban: Participants were administered 6 milligram (mg) IV loading dose of retosiban over 5 minutes followed by a 6 milligram per hour (mg/hour) continuous infusion of retosiban over 48 hours. Participants with an inadequate response any time after first hour of treatment were administered another 6 mg retosiban loading dose followed by 12 mg/hour continuous infusion for remainder of 48-hour treatment period.
Period: Overall Study
Arm/Group | Placebo | Retosiban
Started | 13 | 12
Treated | 13 | 10
Completed | 13 | 10
Not Completed | 0 | 2
Not completed — Other: Randomized and not treated | 0 | 2

BASELINE CHARACTERISTICS:
Population: Maternal intent-to-treat (ITT) Population comprised of all mothers randomly assigned to treatment who have been exposed to study treatment irrespective of their compliance to the planned course of treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Retosiban | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.5 (6.78) | 27.7 (6.73) | 27.0 (6.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 2 | 2 | 4
  Asian-Central/South Asian Heritage | 0 | 1 | 1
  Asian-East Asian Heritage | 1 | 0 | 1
  Asian-Japanese Heritage | 4 | 2 | 6
  Asian-South East Asian Heritage | 1 | 0 | 1
  White-White/Caucasian/European Heritage | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Time to Delivery or Treatment Failure, Whichever Occurs First
Description: Time to delivery or treatment failure is the number of days from the first dose of study treatment until delivery or treatment failure whichever occurs first. Treatment failure is defined as the administration of any putative tocolytic medication for treatment of preterm labor or as prophylaxis of preterm labor. Maternal intent-to-treat (ITT) Population comprised of all mothers randomly assigned to treatment who have been exposed to study treatment irrespective of their compliance to the planned course of treatment. The mean number of days to delivery or treatment failure along with standard deviation has been presented. Statistical analysis was not performed due to early termination of the study and resultant small sample size.
Time Frame: Up to 17 weeks
Population: Maternal ITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Days | 11.10 (14.987) | 18.91 (22.993)

2. Primary Outcome: Number of Neonates With Any Diagnosis From the Neonatal Morbidity and Mortality Composite Component
Description: The neonatal composite endpoint was determined from review of medical records and included the following components: fetal or neonatal death, respiratory distress syndrome (RDS), bronchopulmonary dysplasia, necrotizing enterocolitis or isolated perforation, sepsis based on positive blood culture with clinical features of sepsis, meningitis based on positive results for cerebrospinal fluid culture performed as part of infection workup, retinopathy of prematurity, intraventricular hemorrhage (IVH), white matter injury and cerebellar hemorrhage. Neonates with any of the composite component has been presented. Statistical analysis was not performed due to early termination of study and resultant small sample size. Neonatal ITT Population comprised of all neonates whose mothers were the randomized participants who have been exposed to study treatment, that is, mothers from the ITT Population.
Time Frame: Up to 28 days after the estimated date of delivery (EDD) of 40 0/7 weeks
Population: Neonatal ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 4 | 2

3. Secondary Outcome: Time to Delivery
Description: The time to delivery was calculated as the days between the delivery and start time of the study treatment infusion using the formula: Time to delivery (days) = (date and time of delivery minus date and time of start of infusion) divided by (24 multiplied by 60). The mean number of days to delivery along with standard deviation has been presented.
Time Frame: Up to 17 weeks
Population: Maternal ITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Days | 16.32 (18.595) | 19.18 (22.770)

4. Secondary Outcome: Number of Participants With Births Prior to 37 0/7 Weeks Gestation
Description: Gestational age at birth (weeks) is defined as the gestational age when the baby is born. Participants were considered to have delivered prior to 37 0/7 weeks, that is preterm, if the gestational age at birth is less than 37 0/7 weeks. The number of participants who delivered prior to 37 0/7 weeks gestation has been presented.
Time Frame: Up to 13 weeks
Population: Maternal ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 9 | 8

5. Secondary Outcome: Number of Participants With Births at Term
Description: Participants were considered to have delivered at term if the gestational age was >=37 0/7. The number of participants who delivered at term, that is, 37 0/7 to 41 6/7 weeks gestation has been presented.
Time Frame: Up to 17 weeks
Population: Maternal ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 4 | 2

6. Secondary Outcome: Length of Neonatal Hospital Stay
Description: The length of stay was collected from medical records and was calculated as the days between the delivery date and time and discharge date and time.
Time Frame: Up to 28 days post EDD of 40 0/7 weeks gestation
Population: Neonatal ITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Days | 37.50 (34.537) | 26.05 (32.689)

7. Secondary Outcome: Number of Participants With Births Prior to 35 0/7 Weeks Gestation
Description: The number of participants who delivered prior to 35 0/7 weeks gestation has been presented.
Time Frame: Up to 11 weeks
Population: Maternal ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 9 | 7

8. Secondary Outcome: Number of Participants With Births Prior to 32 0/7 Weeks Gestation
Description: The number of participants who delivered prior to 32 0/7 weeks gestation has been presented. Only those maternal participants who were randomized prior to 32 0/7 week's gestation and delivered were included.
Time Frame: Up to 8 weeks
Population: Maternal ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 9 | 6
Participants | 6 | 2

9. Secondary Outcome: Number of Participants With Births Prior to 28 0/7 Weeks Gestation
Description: The number of participants who delivered prior to 28 0/7 weeks gestation has been presented. Only those maternal participants who were randomized prior to 28 0/7 week's gestation and delivered were included.
Time Frame: Up to 4 weeks
Population: Maternal ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 2 | 2
Participants | 2 | 1

10. Secondary Outcome: Number of Participants With Births <=7 Days From the First Study Treatment
Description: The number of participants who delivered in less than or equal to 7 days from first dose of study treatment has been presented.
Time Frame: Up to 7 days
Population: Maternal ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 5 | 5

11. Secondary Outcome: Number of Participants With Births at <=48 Hours From the First Study Treatment
Description: The number of participants who delivered in less than or equal to 48 hours from first dose of study treatment has been presented.
Time Frame: Up to 48 hours
Population: Maternal ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 3 | 3

12. Secondary Outcome: Number of Participants With Births at <=24 Hours From the First Study Treatment
Description: The number of participants who delivered in less than or equal to 24 hours from first dose of study treatment has been presented.
Time Frame: Up to 24 hours
Population: Maternal ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 3 | 1

13. Secondary Outcome: Number of Neonates With Any of the Co-primary Composite Neonatal Morbidity and Mortality, Excluding RDS
Description: The neonatal composite endpoint was determined from review of medical records and included the following components: fetal or neonatal death, RDS, bronchopulmonary dysplasia, necrotizing enterocolitis or isolated perforation, sepsis based on positive blood culture with clinical features of sepsis, meningitis based on positive results for cerebrospinal fluid culture performed as part of infection workup, retinopathy of prematurity, IVH, white matter injury and cerebellar hemorrhage. The number of neonates with any co-primary composite neonatal morbidity and mortality component, excluding RDS has been presented.
Time Frame: Up to 28 weeks after EDD (40 weeks gestation)
Population: Neonatal ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 3 | 0

14. Secondary Outcome: Number of Neonates With Each Individual Component of the Composite Neonatal Morbidity and Mortality
Description: The neonatal composite endpoint was determined from review of medical records and included the following components: fetal or neonatal death, RDS, bronchopulmonary dysplasia, necrotizing enterocolitis or isolated perforation, sepsis based on positive blood culture with clinical features of sepsis, meningitis based on positive results for cerebrospinal fluid culture performed as part of infection workup, retinopathy of prematurity, IVH, white matter injury and cerebellar hemorrhage. The number of neonates with each individual component of the composite component has been presented.
Time Frame: Up to 28 days after the EDD of 40 0/7 weeks
Population: Neonatal ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants
  Fetal Death | 0 | 0
  Neonatal Death | 0 | 0
  RDS | 3 | 2
  Bronchopulmonary dysplasia | 3 | 0
  Necrotizing enterocolitis or Isolated Perforation | 0 | 0
  Sepsis | 0 | 0
  Meningitis | 0 | 0
  Retinopathy of prematurity | 0 | 0
  IVH | 0 | 0
  White Matter Injury | 0 | 0
  Cerebellar Hemorrhage | 0 | 0

15. Secondary Outcome: Number of Neonatal Participants With Admission to a Particular Hospital Unit
Description: Neonatal healthcare resource utilization was collected from review of medical records. The number of neonatal participants who were admitted to a particular hospital unit that is, level III (or higher) intensive neonatal care (NICU), Intensive care unit (ICU), general ward, Level I - Basic Neonatal care, Well born nursery (SCBU) and Level II-Special Care Newborn nursery high dependency (NHDU) has been summarized. Neonatal Safety Population consisted of neonates whose mothers received study treatment.
Time Frame: Up to 28 days post EDD (40 0/7 weeks gestation)
Population: Neonatal Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants
  Level III (or higher) NICU | 5 | 6
  Intensive care unit | 0 | 1
  General Ward | 2 | 2
  Level II-Special Care NHDU | 0 | 1
  Missing | 1 | 0
  Multiple ward type | 5 | 0

16. Secondary Outcome: Length of Stay in Specialized Care Unit
Description: Neonatal healthcare resource utilization was collected from review of medical records. The length of stay in a specialized care unit (NICU or ICU) has been presented for neonatal participants with admission to ICU or NICU.
Time Frame: Up to 28 days post EDD (40 0/7 weeks gestation)
Population: Neonatal Safety Population.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 10 | 7
Days | 40.34 (35.475) | 35.60 (35.308)

17. Secondary Outcome: Number of Newborn Participants With Hospital Readmission
Description: Newborn hospital readmission following hospitalization for birth was collected from the newborn's medical records. The number of newborn participants who had readmission to hospital is presented.
Time Frame: Up to 28 days of EDD (40 0/7 weeks gestation)
Population: Neonatal Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 0 | 0

18. Secondary Outcome: Length of Stay Following Readmission to Hospital
Description: Newborn hospital readmission following hospitalization for birth was collected from the newborn's medical records. Length of stay in hospital following readmission is presented for neonates.
Time Frame: Up to 28 days after EDD (40 0/7 weeks gestation)
Population: Neonatal Safety Population
Measure: Median (Full Range); unit: Days
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Days | 0 [0 to 0] | 0 [0 to 0]

19. Secondary Outcome: Number of Participants With Ambulatory Surgery
Description: Information regarding participants who had ambulatory surgery was collected from the newborn medical records. The number of neonatal participants with ambulatory surgery is presented.
Time Frame: Up to 28 days post EDD (40 0/7 weeks gestation)
Population: Neonatal Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 0 | 0

20. Secondary Outcome: Time to Treatment Failure
Description: Treatment failure is defined as the administration of any putative tocolytic medication for treatment of preterm labor or as prophylaxis of preterm labor. Time to treatment failure is the number of days from the first dose of study treatment until treatment failure. The mean number of days to delivery or treatment failure along with standard deviation has been presented. Only those maternal participants with treatment failure were included in the analysis. NA indicates standard deviation could not be calculated as only one participant was analyzed.
Time Frame: Up to 17 weeks
Population: Maternal ITT Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 4 | 1
Days | 1.141 (1.4307) | 0.899 (NA) — Standard deviation could not be calculated as only one participant was analyzed.

21. Secondary Outcome: Number of Participants Who Received Any Putative Tocolytic
Description: A putative tocolytic medication was the medication administered for active preterm labor or as prevention of preterm labor and included calcium channel blockers, nonsteroidal anti-inflammatory drugs, or beta agonists, or magnesium sulfate doses that exceeded prespecified IV loading doses, infusion rates, or total duration of administration.
Time Frame: Up to 17 weeks
Population: Maternal Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 4 | 1

22. Secondary Outcome: Number of Participants With Subsequent Preterm Labor
Description: The participants who had not delivered after 48 hours post-infusion were contacted to determine if they had delivered or experienced any subsequent episodes of preterm labor. A subsequent episode of preterm labor was only recorded if the participant reported it to the Principal Investigator during one of the telephone follow-up calls but did not then go on to immediately deliver. However, if labor started and led to immediate delivery, then the only data collected would be the pre-specified delivery data and thus would not be counted as a subsequent episode of preterm labor. The number of participants who had a subsequent episode of preterm labor after administration of the study treatment has been presented. Maternal Safety Population comprised of all maternal participants randomly assigned to treatment who have been exposed to study treatment.
Time Frame: Up to 11 weeks
Population: Maternal Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 1 | 1

23. Secondary Outcome: Number of Maternal Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; important medical events that mey require medical or surgical intervention to prevent one of the other outcomes described before; is associated with liver injury and impaired liver function. Maternal Safety Population comprised of all mothers randomly assigned to treatment who have been exposed to study treatment. The number of maternal participants who experienced at least one AE and one SAE has been presented.
Time Frame: Up to 6 weeks after delivery
Population: Maternal Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants
  AEs | 6 | 6
  SAEs | 0 | 0

24. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP)
Description: SBP and DBP were measured with participants in a semirecumbent or seated position. SBP and DBP were measured during inpatient randomized treatment phase (15 to 30 minutes, 4 to 8 hours, and 20 to 24 hours after the start of the infusion, at the end of the infusion) and at the post-infusion assessment. Baseline is the last available assessment prior to first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to 9 days
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
millimeter of mercury (mmHg)
  DBP; Day 1: 15 to 30 minutes; n=13, 10 | -3.2 (10.64) | -6.8 (8.22)
  DBP; Day 1: 4 to 8 hours; n=11, 10: number analyzed (Participants) | 11 | 10
  DBP; Day 1: 4 to 8 hours; n=11, 10 | -9.0 (11.31) | -7.0 (10.14)
  DBP; Day 1: 20 to 24 hours; n=10, 8: number analyzed (Participants) | 10 | 8
  DBP; Day 1: 20 to 24 hours; n=10, 8 | -13.1 (11.05) | -6.5 (8.65)
  DBP; Day 2; n=11, 7: number analyzed (Participants) | 11 | 7
  DBP; Day 2; n=11, 7 | -10.2 (11.07) | -4.0 (6.66)
  DBP; Post infusion assessment; n=9, 5: number analyzed (Participants) | 9 | 5
  DBP; Post infusion assessment; n=9, 5 | -6.6 (12.69) | -2.8 (4.76)
  SBP; Day 1: 15 to 30 minutes; n=13, 10 | -0.8 (7.50) | -3.1 (10.40)
  SBP; Day 1: 4 to 8 hours; n=11, 10: number analyzed (Participants) | 11 | 10
  SBP; Day 1: 4 to 8 hours; n=11, 10 | -7.1 (13.09) | -1.3 (9.06)
  SBP; Day 1: 20 to 24 hours; n=10, 8: number analyzed (Participants) | 10 | 8
  SBP; Day 1: 20 to 24 hours; n=10, 8 | -5.2 (12.47) | 2.6 (14.56)
  SBP; Day 2; n=11, 7: number analyzed (Participants) | 11 | 7
  SBP; Day 2; n=11, 7 | -4.5 (11.86) | 0.7 (10.21)
  SBP; Post infusion assessment; n=9, 5: number analyzed (Participants) | 9 | 5
  SBP; Post infusion assessment; n=9, 5 | -9.6 (8.69) | -7.0 (8.22)

25. Secondary Outcome: Change From Baseline in Heart Rate
Description: Heart rate was measured with the participants in a semirecumbent or seated position. Heart rate was measured during inpatient randomized treatment phase (15 to 30 minutes, 4 to 8 hours, and 20 to 24 hours after the start of the infusion, at the end of the infusion) and at the post-infusion assessment. Baseline is the last available assessment prior to first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to 9 days
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
beats per minute
  Day 1: 15 to 30 minutes; n=13, 10 | -5.1 (12.37) | 1.4 (8.13)
  Day 1: 4 to 8 hours; n=11, 10: number analyzed (Participants) | 11 | 10
  Day 1: 4 to 8 hours; n=11, 10 | -2.6 (10.82) | -0.3 (8.12)
  Day 1: 20 to 24 hours; n=9, 8: number analyzed (Participants) | 9 | 8
  Day 1: 20 to 24 hours; n=9, 8 | -4.1 (10.61) | 6.5 (21.64)
  Day 2; n=11, 7: number analyzed (Participants) | 11 | 7
  Day 2; n=11, 7 | -5.6 (15.73) | -3.6 (13.91)
  Post infusion assessment; n=9, 5: number analyzed (Participants) | 9 | 5
  Post infusion assessment; n=9, 5 | -6.1 (17.80) | -3.8 (16.24)

26. Secondary Outcome: Change From Baseline in Temperature
Description: Temperature was measured with the participants in a semirecumbent or seated position. Temperature was measured during inpatient randomized treatment phase (15 to 30 minutes, 4 to 8 hours, and 20 to 24 hours after the start of the infusion, at the end of the infusion) and at the post-infusion assessment. Baseline is the last available assessment prior to first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
degree Celsius
  Day 1: 15 to 30 minutes; n=12, 9: number analyzed (Participants) | 12 | 9
  Day 1: 15 to 30 minutes; n=12, 9 | -0.028 (0.4123) | -0.111 (0.1900)
  Day 1: 4 to 8 hours; n=11, 10: number analyzed (Participants) | 11 | 10
  Day 1: 4 to 8 hours; n=11, 10 | 0.087 (0.3947) | -0.144 (0.3594)
  Day 1: 20 to 24 hours; n=10, 8: number analyzed (Participants) | 10 | 8
  Day 1: 20 to 24 hours; n=10, 8 | 0.104 (0.5413) | -0.043 (0.3174)
  Day 2; n=11, 7: number analyzed (Participants) | 11 | 7
  Day 2; n=11, 7 | 0.105 (0.5067) | 0.051 (0.2062)
  Post-infusion assessment; n=9, 5: number analyzed (Participants) | 9 | 5
  Post-infusion assessment; n=9, 5 | -0.136 (0.4668) | 0.072 (0.2234)

27. Secondary Outcome: Change From Baseline in Respiratory Rate
Description: Respiratory rate was measured with the participants in a semirecumbent or seated position. Respiratory rate was measured during inpatient randomized treatment phase (15 to 30 minutes, 4 to 8 hours, and 20 to 24 hours after the start of the infusion, at the end of the infusion) and at the post-infusion assessment. Baseline is the last available assessment prior to first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
breaths per minute
  Day 1: 15 to 30 minutes; n=11, 8: number analyzed (Participants) | 11 | 8
  Day 1: 15 to 30 minutes; n=11, 8 | 0.5 (3.45) | -1.1 (2.90)
  Day 1: 4 to 8 hours; n=8, 9: number analyzed (Participants) | 8 | 9
  Day 1: 4 to 8 hours; n=8, 9 | 1.1 (3.83) | -1.1 (2.15)
  Day 1: 20 to 24 hours; n=9, 7: number analyzed (Participants) | 9 | 7
  Day 1: 20 to 24 hours; n=9, 7 | 0.3 (2.35) | -1.0 (2.77)
  Day 2; n=10, 6: number analyzed (Participants) | 10 | 6
  Day 2; n=10, 6 | 0.9 (4.01) | 0.0 (1.79)
  Post infusion assessment; n=8, 4: number analyzed (Participants) | 8 | 4
  Post infusion assessment; n=8, 4 | 0.4 (4.27) | 0.5 (2.52)

28. Secondary Outcome: Change From Baseline in Hematocrit Levels
Description: Blood samples were collected for the evaluation of change in hematocrit levels from Baseline. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Proportion of red blood cells in blood
  Day 2; n=9, 3: number analyzed (Participants) | 9 | 3
  Day 2; n=9, 3 | -0.0343 (0.04324) | -0.0470 (0.02773)
  Post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  Post-infusion assessment; n=7, 5 | -0.0090 (0.02900) | -0.0078 (0.02928)

29. Secondary Outcome: Change From Baseline in Hemoglobin and Erythrocyte Mean Corpuscular Hemoglobin Concentration (MCHC)
Description: Blood samples were collected for the evaluation of change in hemoglobin levels and MCHC from Baseline. Baseline is defined as the last available assessment prior to the first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
grams per liter (g/L)
  Hemoglobin; Day 2; n=9, 3: number analyzed (Participants) | 9 | 3
  Hemoglobin; Day 2; n=9, 3 | -11.2 (11.20) | -15.7 (6.66)
  Hemoglobin; Post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  Hemoglobin; Post-infusion assessment; n=7, 5 | -1.0 (9.76) | -1.6 (8.79)
  MCHC; Day 2; n=9, 3: number analyzed (Participants) | 9 | 3
  MCHC; Day 2; n=9, 3 | -0.3 (17.27) | -2.7 (10.97)
  MCHC; Post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  MCHC; Post-infusion assessment; n=7, 5 | 5.0 (8.52) | 2.6 (5.41)

30. Secondary Outcome: Change From Baseline in Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Platelets and Leukocytes Count
Description: Blood samples were collected for the evaluation of change in basophils, eosinophils, lymphocytes, monocytes, neutrophils, platelets and leukocytes count. Baseline is defined as the last available assessment prior to the first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: Billion cells per liter (L)
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Billion cells per liter (L)
  Basophils; Day 2; n=9, 3: number analyzed (Participants) | 9 | 3
  Basophils; Day 2; n=9, 3 | -0.003 (0.0132) | 0.000 (0.0458)
  Basophils; post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  Basophils; post-infusion assessment; n=7, 5 | 0.003 (0.0160) | 0.058 (0.1103)
  Eosinophils; Day 2; n=9, 3: number analyzed (Participants) | 9 | 3
  Eosinophils; Day 2; n=9, 3 | 0.004 (0.0938) | -0.063 (0.0513)
  Eosinophils; post-infusion assessment; 7, 5: number analyzed (Participants) | 7 | 5
  Eosinophils; post-infusion assessment; 7, 5 | 0.064 (0.1321) | -0.044 (0.1328)
  Lymphocytes; Day 2; n=9, 3: number analyzed (Participants) | 9 | 3
  Lymphocytes; Day 2; n=9, 3 | 0.323 (0.6117) | 0.877 (0.1914)
  Lymphocytes; post-infusion assessment; 7, 5: number analyzed (Participants) | 7 | 5
  Lymphocytes; post-infusion assessment; 7, 5 | 0.253 (1.0579) | 1.006 (1.4223)
  Monocytes; Day 2; n=9, 3: number analyzed (Participants) | 9 | 3
  Monocytes; Day 2; n=9, 3 | 0.008 (0.3389) | 0.147 (0.5773)
  Monocytes; post-infusion assessment; 7, 5: number analyzed (Participants) | 7 | 5
  Monocytes; post-infusion assessment; 7, 5 | 0.141 (0.2535) | -0.082 (0.4135)
  Neutrophils; Day 2; n=9, 3: number analyzed (Participants) | 9 | 3
  Neutrophils; Day 2; n=9, 3 | 2.744 (6.9362) | -1.813 (3.3001)
  Neutrophils; post-infusion assessment; 7, 5: number analyzed (Participants) | 7 | 5
  Neutrophils; post-infusion assessment; 7, 5 | -2.246 (6.0323) | -1.910 (2.8497)
  Platelets; Day 2; n=8, 3: number analyzed (Participants) | 8 | 3
  Platelets; Day 2; n=8, 3 | -6.4 (47.42) | -24.7 (32.58)
  Platelets; post-infusion assessment; 6, 5: number analyzed (Participants) | 6 | 5
  Platelets; post-infusion assessment; 6, 5 | -15.7 (60.48) | -5.4 (33.34)
  Leukocytes; Day 2; n=9, 3: number analyzed (Participants) | 9 | 3
  Leukocytes; Day 2; n=9, 3 | 3.10 (6.720) | -0.87 (2.914)
  Leukocytes; post-infusion assessment; 7, 5: number analyzed (Participants) | 7 | 5
  Leukocytes; post-infusion assessment; 7, 5 | -1.76 (5.358) | -0.98 (2.645)

31. Secondary Outcome: Change From Baseline in Erythrocyte Mean Corpuscular Volume (MCV) and Mean Platelet Volume (MPV)
Description: Blood samples were collected for the evaluation of change in MCV and MPV from Baseline. Baseline is defined as the last available assessment prior to the first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: femtoliter (fL)
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
femtoliter (fL)
  MCV; Day 2; n=9, 3: number analyzed (Participants) | 9 | 3
  MCV; Day 2; n=9, 3 | 0.4 (2.79) | 1.7 (4.73)
  MCV; Post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  MCV; Post-infusion assessment; n=7, 5 | -1.9 (1.77) | -0.8 (1.30)
  MPV; Day 2; n=8, 3: number analyzed (Participants) | 8 | 3
  MPV; Day 2; n=8, 3 | -0.11 (0.455) | -0.20 (0.436)
  MPV; Post-infusion assessment; n=6, 5: number analyzed (Participants) | 6 | 5
  MPV; Post-infusion assessment; n=6, 5 | 0.02 (0.833) | 0.48 (1.026)

32. Secondary Outcome: Change From Baseline in Erythrocyte Level
Description: Blood samples were collected for the evaluation of change in erythrocyte level from Baseline. Baseline is defined as the last available assessment prior to the first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: Trillion cells per liter
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Trillion cells per liter
  Day 2; n=9, 3: number analyzed (Participants) | 9 | 3
  Day 2; n=9, 3 | -0.39 (0.423) | -0.53 (0.153)
  Post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  Post-infusion assessment; n=7, 5 | -0.03 (0.330) | -0.02 (0.303)

33. Secondary Outcome: Change From Baseline in Alkaline Phosphatase (ALP), Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Gamma Glutamyl Transferase (GGT) and Lactate Dehydrogenase (LDH) Levels
Description: Blood samples were collected for the evaluation of change in ALP, ALT, AST, GGT and LDH from Baseline. Baseline is defined as the last available assessment prior to the first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: International Units per liter (IU/L)
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
International Units per liter (IU/L)
  ALP; Day 2; n=9, 5: number analyzed (Participants) | 9 | 5
  ALP; Day 2; n=9, 5 | -17.3 (17.56) | -11.8 (6.46)
  ALP; post-infusion assessment; n=8, 6: number analyzed (Participants) | 8 | 6
  ALP; post-infusion assessment; n=8, 6 | 6.6 (31.14) | -2.8 (14.08)
  ALT; Day 2; n=9, 5: number analyzed (Participants) | 9 | 5
  ALT; Day 2; n=9, 5 | 3.9 (19.60) | 4.4 (10.64)
  ALT; post-infusion assessment; n=8, 6: number analyzed (Participants) | 8 | 6
  ALT; post-infusion assessment; n=8, 6 | -8.8 (20.04) | 2.5 (5.50)
  AST; Day 2; n=9, 5: number analyzed (Participants) | 9 | 5
  AST; Day 2; n=9, 5 | 4.4 (15.69) | 2.0 (10.20)
  AST; post-infusion assessment; n=8, 6: number analyzed (Participants) | 8 | 6
  AST; post-infusion assessment; n=8, 6 | -9.1 (13.05) | -0.5 (7.45)
  GGT; Day 2; n=9, 5: number analyzed (Participants) | 9 | 5
  GGT; Day 2; n=9, 5 | -0.9 (1.69) | -0.8 (1.30)
  GGT; post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  GGT; post-infusion assessment; n=7, 5 | 4.4 (2.57) | 0.4 (2.07)
  LDH; Day 2; n=9, 5: number analyzed (Participants) | 9 | 5
  LDH; Day 2; n=9, 5 | -6.7 (33.51) | -26.4 (31.86)
  LDH; post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  LDH; post-infusion assessment; n=7, 5 | -8.1 (21.93) | -7.6 (31.76)

34. Secondary Outcome: Change From Baseline in Albumin and Protein Levels
Description: Blood samples were collected for the evaluation of change in albumin and protein levels from Baseline. Baseline is defined as the last available assessment prior to the first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
grams per liter (g/L)
  Albumin; Day 2; n=9, 5: number analyzed (Participants) | 9 | 5
  Albumin; Day 2; n=9, 5 | -3.4 (3.68) | -2.6 (1.67)
  Albumin; post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  Albumin; post-infusion assessment; n=7, 5 | -1.3 (2.21) | -1.0 (2.35)
  Protein; Day 2; n=9, 5: number analyzed (Participants) | 9 | 5
  Protein; Day 2; n=9, 5 | -5.8 (6.26) | -5.4 (3.58)
  Protein; post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  Protein; post-infusion assessment; n=7, 5 | -2.4 (3.41) | -1.8 (5.02)

35. Secondary Outcome: Change From Baseline in Anion Gap, Calcium, Chloride, Carbon Dioxide, Glucose, Potassium, Magnesium, Phosphate and Sodium Level
Description: Blood samples were collected for the evaluation of change from Baseline in levels of anion gap, calcium, chloride, carbon dioxide, glucose, potassium, magnesium, phosphate, and sodium. Baseline is defined as the last available assessment prior to the first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
millimoles per liter (mmol/L)
  Anion Gap; Day 2; n=8, 4: number analyzed (Participants) | 8 | 4
  Anion Gap; Day 2; n=8, 4 | 0.0 (4.72) | 0.0 (1.83)
  Anion Gap; post-infusion assessment; n=7, 4: number analyzed (Participants) | 7 | 4
  Anion Gap; post-infusion assessment; n=7, 4 | -1.6 (5.26) | 0.3 (2.22)
  Calcium; Day 2; n=9, 5: number analyzed (Participants) | 9 | 5
  Calcium; Day 2; n=9, 5 | -0.042 (0.2833) | -0.040 (0.1208)
  Calcium; post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  Calcium; post-infusion assessment; n=7, 5 | 0.091 (0.2052) | -0.048 (0.1016)
  Chloride; Day 2; n=9, 5: number analyzed (Participants) | 9 | 5
  Chloride; Day 2; n=9, 5 | 1.0 (5.17) | 1.8 (2.17)
  Chloride; post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  Chloride; post-infusion assessment; n=7, 5 | -0.7 (3.35) | -0.6 (2.30)
  Carbon Dioxide; Day 2; n=9, 5: number analyzed (Participants) | 9 | 5
  Carbon Dioxide; Day 2; n=9, 5 | -0.2 (3.63) | 0.0 (2.35)
  Carbon Dioxide; post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  Carbon Dioxide; post-infusion assessment; n=7, 5 | 2.3 (3.64) | -0.2 (2.77)
  Glucose; Day 2; n=9, 5: number analyzed (Participants) | 9 | 5
  Glucose; Day 2; n=9, 5 | 1.47 (1.639) | 1.98 (1.064)
  Glucose; post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  Glucose; post-infusion assessment; n=7, 5 | 0.11 (2.497) | 0.28 (2.109)
  Potassium; Day 2; n=9, 5: number analyzed (Participants) | 9 | 5
  Potassium; Day 2; n=9, 5 | -0.16 (0.394) | 0.10 (0.515)
  Potassium; post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  Potassium; post-infusion assessment; n=7, 5 | -0.16 (0.237) | 0.10 (0.283)
  Magnesium; Day 2; n=9, 5: number analyzed (Participants) | 9 | 5
  Magnesium; Day 2; n=9, 5 | -0.411 (0.9476) | -0.236 (0.5428)
  Magnesium; post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  Magnesium; post-infusion assessment; n=7, 5 | -0.449 (0.6473) | -0.056 (0.6199)
  Phosphate; Day 2; n=9, 5: number analyzed (Participants) | 9 | 5
  Phosphate; Day 2; n=9, 5 | -0.133 (0.1768) | 0.030 (0.2928)
  Phosphate; post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  Phosphate; post-infusion assessment; n=7, 5 | 0.021 (0.2018) | 0.110 (0.1557)
  Sodium; Day 2; n=9, 5: number analyzed (Participants) | 9 | 5
  Sodium; Day 2; n=9, 5 | 1.4 (2.96) | 0.4 (1.67)
  Sodium; post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  Sodium; post-infusion assessment; n=7, 5 | 0.1 (2.12) | -0.8 (1.64)

36. Secondary Outcome: Change From Baseline in Direct Bilirubin, Bilirubin, Indirect Bilirubin, Creatinine and Urate Levels
Description: Blood samples were collected for the evaluation of change from Baseline in levels of direct bilirubin, bilirubin, indirect bilirubin, creatinine and urate. Baseline is defined as the last available assessment prior to the first dose of study treatment. Change from Baseline is the post-dose visit value minus Baseline. Only those participants with data available at the specified data points were analyzed (represented by n=X in category title).
Time Frame: Baseline and up to 1 week
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: micromoles per liter (µmol/L)
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
micromoles per liter (µmol/L)
  Direct Bilirubin; Day 2; n=9, 5: number analyzed (Participants) | 9 | 5
  Direct Bilirubin; Day 2; n=9, 5 | 0.0 (1.00) | -0.4 (0.89)
  Direct Bilirubin; post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  Direct Bilirubin; post-infusion assessment; n=7, 5 | 0.3 (0.76) | -0.4 (0.89)
  Bilirubin; Day 2; n=9, 5: number analyzed (Participants) | 9 | 5
  Bilirubin; Day 2; n=9, 5 | -0.7 (1.41) | -0.8 (1.10)
  Bilirubin; post-infusion assessment; n=8, 6: number analyzed (Participants) | 8 | 6
  Bilirubin; post-infusion assessment; n=8, 6 | -0.3 (1.28) | -2.0 (3.10)
  Indirect Bilirubin; Day 2; n=9, 5: number analyzed (Participants) | 9 | 5
  Indirect Bilirubin; Day 2; n=9, 5 | -0.7 (1.41) | -0.4 (1.67)
  Indirect Bilirubin; post-infusion assessment;n=7,5: number analyzed (Participants) | 7 | 5
  Indirect Bilirubin; post-infusion assessment;n=7,5 | -0.6 (1.51) | -1.6 (3.85)
  Creatinine; Day 2; n=6, 3: number analyzed (Participants) | 6 | 3
  Creatinine; Day 2; n=6, 3 | -0.33 (6.812) | 2.37 (1.429)
  Creatinine; post-infusion assessment; n=6, 3: number analyzed (Participants) | 6 | 3
  Creatinine; post-infusion assessment; n=6, 3 | 1.92 (5.075) | -0.33 (2.695)
  Urate; Day 2; n=9, 5: number analyzed (Participants) | 9 | 5
  Urate; Day 2; n=9, 5 | 1.1 (24.72) | -22.0 (13.04)
  Urate; post-infusion assessment; n=7, 5: number analyzed (Participants) | 7 | 5
  Urate; post-infusion assessment; n=7, 5 | 12.9 (24.30) | -2.0 (40.25)

37. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due to Clinical and Laboratory Toxicities
Description: Number of maternal participants who discontinued study treatment due to clinical and laboratory toxicities is presented.
Time Frame: Up to 48 hours post-infusion
Population: Maternal Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 0 | 0

38. Secondary Outcome: Number of Maternal Participants With a Score of 12 or Higher on the Edinburgh Postnatal Depression Scale (EPDS)
Description: The effect of preterm birth on maternal health status was assessed using the EPDS. The EPDS is a 10-item self-reported assessment of depression, validated for administration during both the antenatal and the post-natal periods. Items are rated on a 4-point variable Likert scale, ranging from 0 to 3. The total score was calculated by adding individual scores for each item and ranged from 0 to 30. A score of less than 8 indicates depression not likely; score of 9 to 11 indicates possible depression and a score of more than 12 indicates an increased probability of depression. Maternal participants were required to complete the EPDS at the maternal follow-up assessment 6 weeks post-delivery.
Time Frame: Up to 6 weeks post delivery
Population: Maternal Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 2 | 0

39. Secondary Outcome: Number of Maternal Participants With AEs of Special Interest (AESI).
Description: Maternal AESI included: maternal death; chorioamnionitis and its complications (clinical chorioamnionitis, preterm premature rupture of membranes, endomyometritis, wound infection, pelvic abscess, bacteremia, septic shock, disseminated intravascular coagulation, and adult RDS); placental abruption; postpartum hemorrhage - postpartum hemorrhage and/or retained placenta and pulmonary edema. The number of participants with at least one AESI has been presented.
Time Frame: Up to 6 weeks post-delivery
Population: Maternal Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 0 | 1

40. Secondary Outcome: Number of Maternal Participants With Disease Related AEs (DRE)
Description: Maternal DREs included: signs and symptoms of labor discomfort (example, cramping, backache, muscle aches, nausea); subsequent episodes of preterm labor and hospitalization for delivery. The number of participants with at least one DRE has been presented.
Time Frame: Up to 6 weeks post-delivery
Population: Maternal Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 0 | 1

41. Secondary Outcome: Number of Fetal Participants With AEs and SAEs Prior to Delivery
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; important medical events that may require medical or surgical intervention to prevent one of the other outcomes described before; is associated with liver injury and impaired liver function. Fetal AEs and SAEs included the adverse events that were experienced by the fetus prior to delivery. The number of fetal participants who experienced at least one AE and one SAE has been presented.
Time Frame: Up to 17 weeks post-infusion
Population: Maternal Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants
  AE | 3 | 5
  SAE | 0 | 1

42. Secondary Outcome: Number of Participants With Fetal Acidosis
Description: The number of participants with fetal acidosis is presented.
Time Frame: Up to 16 weeks
Population: Maternal Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 0 | 0

43. Secondary Outcome: Number of Participants With Fetal AESI
Description: Fetal AESI included: intrauterine fetal demise; category II or III fetal heart rate tracing; and fetal inflammatory response syndrome characterized by cord blood interleukin-6 >11 picogram per milliliter (pg/mL), funisitis, or chorionic vasculitis. The number of participants who experienced at least one AESI has been presented.
Time Frame: Up to 17 weeks
Population: Maternal Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 3 | 5

44. Secondary Outcome: Neonatal APGAR Scores
Description: APGAR is a quick test to assess the health of new born children. The test is performed at 1 and 5 minutes after birth. APGAR scale is determined by evaluating the new born on five categories (appearance, pulse, grimace, activity and respiration) on a scale from zero to two, then summing up the five values obtained. APGAR score ranges from 0 to 10 where a score of 7 and above is normal. The mean and standard deviation of APGAR scores at one minute and at five minutes of birth has been presented.
Time Frame: Up to 5 minutes after birth
Population: Neonatal ITT Population
Measure: Mean (Standard Deviation); unit: Score on APGAR scale
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Score on APGAR scale
  one minute at birth | 7.3 (1.80) | 7.5 (1.78)
  five minutes at birth | 8.5 (1.05) | 8.7 (1.06)

45. Secondary Outcome: Weight of Neonates
Description: The weight of neonates was obtained from the neonate birth record. The mean weight of neonates and standard deviation has been presented.
Time Frame: Up to 17 weeks
Population: Neonatal ITT Population
Measure: Mean (Standard Deviation); unit: grams (g)
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
grams (g) | 2015.0 (805.67) | 2121.2 (681.31)

46. Secondary Outcome: Head Circumference of Neonates
Description: The head circumference was determined from the neonate birth record.
Time Frame: Up to 17 weeks
Population: Neonatal ITT Population
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
centimeters (cm) | 29.57 (2.791) | 30.13 (3.059)

47. Secondary Outcome: Number of Neonatal Participants With AEs and SAEs
Description: An AE is any untoward medical occurrence in a clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose: results in death; is life threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect; important medical events that may require medical or surgical intervention to prevent one of the other outcomes described before; is associated with liver injury and impaired liver function. The number of participants who experienced at least one AE and one SAE has been presented. Neonatal Safety Population consisted of neonates whose mothers received randomized treatment.
Time Frame: Up to 28 days after the EDD of 40 weeks gestation
Population: Neonatal Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants
  AEs | 8 | 7
  SAEs | 3 | 5

48. Secondary Outcome: Number of Neonatal Participants With AESI
Description: Neonatal AESI included: Neonatal death; Asphyxia; Infections (early onset neonatal sepsis, septic shock, pneumonia, meningitis); RDS; Hypotension; IVH/periventricular leukomalacia; Bronchopulmonary dysplasia; Neonatal acidosis; Hyperbilirubinemia; Necrotizing enterocolitis; and Hypoxic ischemic encephalopathy. The number of neonatal participants who experienced at least one AESI has been presented.
Time Frame: Up to 28 days after EDD of 40 weeks gestation
Population: Neonatal Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 8 | 5

49. Secondary Outcome: Number of Neonatal Participants With DRE
Description: The disease related neonatal events occurring in Infants born prior to 37 completed weeks included: apnea (severe), respiratory failure due to fatigue, hypoxia, or air leak from alveolar injury, patent ductus arteriosus, bradycardia, ventriculomegaly, cerebellar hemorrhage, hydrocephalus other than congenital, gastroesophageal reflux, aspiration pneumonia, anemia, retinopathy of prematurity (all stages), hearing disorder, temperature instability and hypoglycemia. The number of participants with at least one DRE has been presented.
Time Frame: Up to 28 days after EDD of 40 weeks gestation
Population: Neonatal Safety Population
Measure: Number; unit: Participants
Groups:
- Placebo: Placebo was 0.9 percent sodium chloride infusion matched for retosiban volume, intravenous (IV) loading dose over 5 minutes and continuous infusion rate for remainder of 48-hour treatment period.Placebo was 0.9 percent sodium chloride infusion matched for retosiban volume, IV loading dose over 5 minutes and continuous infusion rate including dose increase in participants with an inadequate response any time after first hour of treatment.
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants | 4 | 2

50. Secondary Outcome: Maternal Length of Stay in Hospital
Description: Details on maternal health care resource use (both for hospitalizations related to preterm labor not resulting in a delivery and hospitalizations related to preterm labor/normal labor resulting in a delivery) associated with an episode of preterm labor, preterm delivery and normal term delivery (>= 37 weeks gestation) were collected from review of medical records. Length of hospital stay associated with hospital admission for preterm labor and normal term labor/term delivery is presented. One participant in the retosiban arm did not have hospitalization data; hence, was excluded from the analysis at delivery. Only participants with data available at the specified time points were analyzed (indicated by n=X) in category titles. NA indicates standard deviation could not be calculated as only one participant was analyzed.
Time Frame: Up to 28 days post EDD (40 0/7 weeks gestation)
Population: Maternal Safety Population
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Days
  Preterm labor; n=1, 0: number analyzed (Participants) | 1 | 0
  Preterm labor; n=1, 0 | 2.642 (NA) — Standard deviation could not be calculated as only one participant was analyzed. |
  Preterm delivery; n=9, 7: number analyzed (Participants) | 9 | 7
  Preterm delivery; n=9, 7 | 10.177 (11.9312) | 13.583 (20.7670)
  Normal term delivery; n=4, 2: number analyzed (Participants) | 4 | 2
  Normal term delivery; n=4, 2 | 3.719 (2.2309) | 4.635 (2.7616)

51. Secondary Outcome: Number of Participants With Hospital Admissions Related to Preterm Labor and Preterm Delivery
Description: Maternal healthcare resource utilization associated with an episode of preterm labor and preterm delivery were collected from the review of medical records. One participant in the retosiban arm did not have hospitalization data; hence, was excluded from the analysis at delivery. The number of participants who had hospital admission for preterm labor and preterm delivery has been presented. Only those participants with data available at the specified time points were analyzed (indicated by n=X in category titles).
Time Frame: Up to 28 days after EDD (40 0/7 weeks of gestation)
Population: Maternal Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants
  Preterm labor; n=13, 10 | 1 | 0
  Preterm delivery; n=13, 9: number analyzed (Participants) | 13 | 9
  Preterm delivery; n=13, 9 | 9 | 7

52. Secondary Outcome: Number of Participants Admitted to Particular Hospital Unit
Description: Maternal healthcare resource utilization associated with an episode of preterm labor, preterm delivery and normal term delivery were collected from the review of medical records. The number of participants who were admitted to a particular hospital unit has been presented.
Time Frame: Up to 28 days post EDD (40 0/7 weeks gestation)
Population: Maternal Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants
  General ward | 9 | 2
  Private/Semi-private room | 3 | 2
  Labor and delivery | 2 | 3
  Labor and delivery to post-partum | 0 | 1
  Post-partum | 0 | 1
  Ward not specified | 0 | 1
  Labor ward | 0 | 1
  Antenatal ward | 0 | 1
  Postnatal ward | 0 | 1

53. Secondary Outcome: Number of Participants With Different Modes of Transportation to Hospital
Description: The means by which the maternal participants were transported to the hospital i.e. ground ambulance/emergency vehicle (gr. amb/emer. veh), air ambulance, family member or other means were obtained from the review of medical records. The number of maternal participants with the corresponding mode of transportation is presented for preterm labor visit and delivery visit. Only those participants with data available at specified time points were analyzed (indicated by n=X in category titles).
Time Frame: Up to 28 days post EDD (40 0/7 weeks gestation)
Population: Maternal Safety Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Retosiban
Number analyzed (Participants) | 13 | 10
Participants
  Preterm labor; gr. amb/emer. veh; n=1, 0: number analyzed (Participants) | 1 | 0
  Preterm labor; gr. amb/emer. veh; n=1, 0 | 0 |
  Preterm labor; air ambulance; n=1, 0: number analyzed (Participants) | 1 | 0
  Preterm labor; air ambulance; n=1, 0 | 0 |
  Preterm labor; family member; n=1, 0: number analyzed (Participants) | 1 | 0
  Preterm labor; family member; n=1, 0 | 1 |
  Preterm labor; other; n=1, 0: number analyzed (Participants) | 1 | 0
  Preterm labor; other; n=1, 0 | 0 |
  Delivery; gr. amb/emer. veh; n=5, 5: number analyzed (Participants) | 5 | 5
  Delivery; gr. amb/emer. veh; n=5, 5 | 2 | 1
  Delivery; air ambulance; n=5, 5: number analyzed (Participants) | 5 | 5
  Delivery; air ambulance; n=5, 5 | 0 | 0
  Delivery; family member; n=5, 5: number analyzed (Participants) | 5 | 5
  Delivery; family member; n=5, 5 | 3 | 3
  Delivery; other; n=5, 5: number analyzed (Participants) | 5 | 5
  Delivery; other; n=5, 5 | 0 | 1
  Preterm labor;<24 hour stay;gr. amb/emer.veh;n=1,0: number analyzed (Participants) | 1 | 0
  Preterm labor;<24 hour stay;gr. amb/emer.veh;n=1,0 | 0 |
  Preterm labor; <24 hour stay;air ambulance; n=1, 0: number analyzed (Participants) | 1 | 0
  Preterm labor; <24 hour stay;air ambulance; n=1, 0 | 0 |
  Preterm labor; <24 hour stay;family member; n=1, 0: number analyzed (Participants) | 1 | 0
  Preterm labor; <24 hour stay;family member; n=1, 0 | 1 |
  Preterm labor; <24 hour stay;other; n=1, 0: number analyzed (Participants) | 1 | 0
  Preterm labor; <24 hour stay;other; n=1, 0 | 0 |

54. Secondary Outcome: Retosiban Clearance
Description: Maternal blood samples were collected at the indicated time points for pharmacokinetic analysis. Data is a combined data set. Data is presented for 10 participants from retosiban arm of study 200719 (NCT02377466) and 43 participants from retosiban arm of study 200721 (NCT02292771).
Time Frame: Day 1 (2 to 4 hours, 10 to 14 hours) and Day 2 (22 to 26 hours, and 48 to 54 hours) post-infusion
Population: Maternal Safety Population. Data is a combined data set. Data is presented for 10 participants from retosiban arm of study 200719 (NCT02377466) and 43 participants from retosiban arm of study 200721 (NCT02292771).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour
Arm/Group | Retosiban
Number analyzed (Participants) | 53
Liters per hour | 83.4 (5.25)

55. Secondary Outcome: Volume of Distribution of Retosiban
Description: as for outcome 54
Time Frame: Day 1 (2 to 4 hours, 10 to 14 hours) and Day 2 (22 to 26 hours, and 48 to 54 hours) post-infusion
Population: as for outcome 54
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Retosiban
Number analyzed (Participants) | 53
Liters | 68.6 (109)

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) will be collected from the start of study treatment and until the follow up contact (Up to 6 weeks after delivery).
Description: SAEs and AEs were analyzed in Maternal Safety Population and Neonatal Safety Population which comprised of mothers randomly assigned to treatment who were exposed to study treatment and neonates whose mothers received randomized treatment.
Groups:
- Placebo (Maternal); Placebo (Fetal); Placebo (Neonatal): Placebo was 0.9 percent sodium chloride infusion matched for retosiban volume, IV loading dose over 5 minutes and continuous infusion rate including dose increase in participants with an inadequate response any time after first hour of treatment.
- Retosiban (Maternal); Retosiban (Fetal); Retosiban (Neonatal): Participants were administered 6 milligram (mg) IV loading dose of retosiban over 5 minutes followed by a 6 milligram per hour (mg/hour) continuous infusion of retosiban over 48 hours. Participants with an inadequate response any time after first hour of treatment were administered another 6 mg retosiban loading dose followed by 12 mg/hour continuous infusion for remainder of 48-hour treatment period.
Arm/Group | Placebo (Maternal) | Retosiban (Maternal) | Placebo (Fetal) | Retosiban (Fetal) | Placebo (Neonatal) | Retosiban (Neonatal)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10 | 0/13 | 0/10 | 0/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/10 | 0/13 | 1/10 | 3/13 | 5/10
Other Adverse Events (participants affected / at risk) | 6/13 | 6/10 | 3/13 | 5/10 | 8/13 | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Maternal) (N=13) | Retosiban (Maternal) (N=10) | Placebo (Fetal) (N=13) | Retosiban (Fetal) (N=10) | Placebo (Neonatal) (N=13) | Retosiban (Neonatal) (N=10)
Umbilical cord prolapse (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Meconium plug syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1
Ankyloglossia congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1
Congenital hypothyroidism (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Group B streptococcus neonatal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tracheitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Selective eating disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Maternal) (N=13) | Retosiban (Maternal) (N=10) | Placebo (Fetal) (N=13) | Retosiban (Fetal) (N=10) | Placebo (Neonatal) (N=13) | Retosiban (Neonatal) (N=10)
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Amniotic cavity infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Bacterial vulvovaginitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Blood calcium decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Uterine contractions abnormal (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Foetal heart rate disorder (Cardiac disorders) | 0 | 0 | 2 | 5 | 0 | 0
Foetal heart rate deceleration abnormality (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 6 | 4
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 2
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Necrotising colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Feeding intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Motor dysfunction (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Intertrigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Granuloma (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Body temperature fluctuation (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-09-08): https://cdn.clinicaltrials.gov/large-docs/66/NCT02377466/SAP_000.pdf
  • Study Protocol (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT02377466/Prot_001.pdf